CLINICAL TRIAL: NCT06817460
Title: A Single Center, Randomized, Single Blind, Parallel Controlled Clinical Study Comparing the Effectiveness and Safety of Three Surgical Pathways for Laparoscopic Total Hysterectomy
Brief Title: A Clinical Study Comparing the Effectiveness and Safety of Three Surgical Pathways for Laparoscopic Total Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024105
Record Dates: First submitted 2024-04-21; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Benign Tumor of Uterus; Surgical Approaches; Enhanced Recovery After Surgery
Keywords: hysterectomy; single-port; multi-port; enhanced recovery after surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Observation group1 (Experimental): tran-sumbilical laparoendoscopic single-site surgery
  Interventions: Procedure: tran-sumbilical laparoendoscopic single-site surgery
- Observation group2 (Experimental): transvaginal natural orifice transluminal endoscopic surgery
  Interventions: Procedure: transvaginal natural orifice transluminal endoscopic surgery
- control group (No Intervention): conventional three-port totaI laparoscopic hysterectomy

INTERVENTIONS:
Procedure: tran-sumbilical laparoendoscopic single-site surgery — Different types of surgery
  Arms: Observation group1
Procedure: transvaginal natural orifice transluminal endoscopic surgery — Different types of surgery
  Arms: Observation group2

SUMMARY:
To explore the achievement of ERAS composite indexes within 24 hours after the operation of transumbilical single-hole laparoscopic total hysterectomy, transvaginal laparoscopic total hysterectomy and porous laparoscopic total hysterectomy.

DETAILED DESCRIPTION:
To explore the achievement of ERAS composite indexes within 24 hours after the operation of transumbilical single-hole laparoscopic total hysterectomy, transvaginal laparoscopic total hysterectomy and porous laparoscopic total hysterectomy.To explore the differences of operation time, intraoperative blood loss, intraoperative conversion mode and postoperative complication rate of three surgical paths: transumbilical single-hole laparoscopic total hysterectomy, transcolposcopic total hysterectomy and porous laparoscopic total hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 females
* Total hysterectomy indications (uterine fibroids, adenomyosis, cervical precancerous lesions, endometrial dysplasia, cervical carcinoma in situ), total hysterectomy is planned
* The patients who participated in the study recognized three surgical paths and were willing to accept any of the three at random
* Be able to understand the research program and voluntarily participate in the research, and sign the informed consent
* Good compliance, able to cooperate with and provide corresponding clinical information
* Complete imaging and pathological clinical data;
* General condition: ECOG≤1; 0 The activity capacity is completely normal, and there is no difference between the activity capacity and that before the onset of the disease; 1 Can move about freely and engage in light physical activity, including general household or office work, but cannot engage in heavy physical activity.

Exclusion Criteria:

* asexual life history
* The cyst needs to be removed at the same time or there are other vulvar, vaginal, appendix and other lesions, and surgical intervention is required at the same time
* Malignant tumors or highly suspected malignant tumors
* History of two or more pelvic surgeries, severe pelvic adhesions(triad examination suspected rectal endometriosis, or poor intrauterine mobility)
* History of peritoneal dialysis, pelvic radiotherapy, and previous history of pelvic laparoscopic tuberculosis
* the uterus is greater than 3 months of pregnancy or the maximum meridian of the uterus is greater than 12cm according to ultrasound (either of the two conditions can be excluded)
* Diabetic patients with unsatisfactory blood sugar control
* BMI>30Kg/m2
* History of severe mental illness and brain dysfunction
* A history of drug abuse or use
* Patients with poor compliance or who are too far away for adequate follow-up

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Achievement of ERAS composite indexes within 24 hours after surgery | (1) 6 hours after surgery; (2) 24 hours after surgery; (3) 48 hours after surgery
  Including: (1) postoperative liquid diet, (2) anal exhaust, (3) self-urination after catheter removal, (4) getting out of bed, (5) visual analogue scale (VAS) score ≤3

SECONDARY OUTCOMES:
Operation time | The operation time is measured in minutes from the beginning of the skin (or vaginal) incision to the completion of the skin (or vaginal) suture
  duration of surgery
intraoperative blood loss | The operation time is measured in minutes from the beginning of the skin (or vaginal) incision to the completion of the skin (or vaginal) suture
  intraoperative blood loss

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China